CLINICAL TRIAL: NCT03741569
Title: Development of a Real-time Signal Processing Algorithm, for Beat-beat Measurement of Fetal Heart Rate and Uterine Contractions by Coupling Non-invasive ABDOminal Sensors
Brief Title: Multisensor Technology for Beat to Beat Fetal Heart Rate Measurement
Acronym: RCF-ABDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017_63; 2018-A01194-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obstetric Labor
Keywords: Fetal heart rate; Multiple sensors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- parturients (gestational age ≥37 weeks). (Other)
  Interventions: Device: Transabdominal Fetal Heart Rate

INTERVENTIONS:
Device: Transabdominal Fetal Heart Rate — Doppler, ECG and acoustic sensors will be placed on the mother's abdomen to capture the heart rate of the fetus and mother as well as uterine contractions.
  For each of the participants, we will make two 15-minute recordings: one with conventional ECG electrodes and one with ECG textile electrodes
  Other Names: Fetal heart rate recording

SUMMARY:
The CIC-IT 1403 laboratory of the University Hospital of Lille has developed a technological solution for acquiring and synchronizing abdominal ECG, acoustic and Doppler signals.

The purpose of this clinical trial is to build a database of signals issued from this device to develop signal processing algorithms to allow optimization of the fetal heart rate calculation.

This study will be carried out in the maternity ward of the Jeanne de Flandre Hospital in the maternal-fetal pathology department Doppler, ECG and acoustic sensors will be placed on the mother's abdomen to capture the heart rate of the fetus and mother as well as uterine contractions.

For each of the participants, we will make two 15-minute recordings: one with conventional ECG electrodes and one with ECG textile electrodes.

This procedure will not affect the usual care of the patient

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Age>18 years

Exclusion Criteria:

* Multiple pregnancy
* Medical termination of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant woman
Enrollment: 90 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
The fetal heart rate signal | at 15 minutes
  The fetal heart rate signal extraction algorithm will be based on the various signal processing tools developed by the INSERM CIC-IT 1403 laboratory

SECONDARY OUTCOMES:
The uterine contraction signal | at 15 minutes
  The uterine contraction signal extraction algorithm will be based on the different signal processing tools developed by the INSERM CIC-IT 1403 laboratory.
Measuring the root mean square deviation between the heart rate signals from the device and the Doppler | at 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Charles Garrabedian, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France